CLINICAL TRIAL: NCT01310647
Title: Prospective Randomized Controlled Trial of Antral Follicle Priming Prior to IVF-ICSI in Previously Diagnosed Low Responders.
Brief Title: Antral Follicle Priming Prior to ICSI (Intracytoplasmic Sperm Injection) in Previously Diagnosed Low Responders
Acronym: FOLLPRIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-018009-26; 2009-018009-26 (EudraCT Number)
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Ovarian Diseases
Keywords: estradiol; testosterone; combined oral contraceptive; low responders; ICSI
MeSH Terms: conditions — Ovarian Diseases | interventions — Testosterone; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Testosterone (Experimental): Transdermal testosterone (20µg/day) from day 24 of the previous cycle until day 2 of the ICSI cycle
  Interventions: Drug: Testosterone
- Estradiol (Experimental): Transdermal estradiol (200µg/day)from day 20 of the previous cycle to day 3 of the ICSI cycle
  Interventions: Drug: Estradiol
- CombEq (Experimental): * (150µg Desogestrel + 30µg Ethinylestradiol)/day during the luteal phase of the two cycles prior to the ICSI
  * Estradiol valerate 4 mg/day during 10 days, starting the second day of the cycle prior to the ICSI cycle.
  Interventions: Drug: CombEq

INTERVENTIONS:
Drug: Testosterone — Transdermal testosterone (20µg/kg/day)from day 24 of the previous cycle to day 2 of the ICSI cycle
  Other Names: Testopatch, Pierre Fabre Ibérica S.A.
  Arms: Testosterone
Drug: Estradiol — Transdermal estradiol (200µg/day)from day 20 of the previous cycle to day 3 of the ICSI cycle
  Other Names: Alcis 100, Chiesi España
  Arms: Estradiol
Drug: CombEq — (150µg Desogestrel + 30µg Ethinylestradiol)/day during the luteal phase of the two cycles prior to the ICSI.
  Valerate estradiol 4mg/day during 10 days, starting the second day of the cycle prios to the ICSI cycle.
  Other Names: Microdiol, MERCK SHARP & DOHME; Meriestra 2mg, Novartis Farmacéutica, S.A.
  Arms: CombEq

SUMMARY:
The aim of this study is to compare the effectiveness of testosterone,estradiol and a combined treatment with estrogens/progestagens prior to IVF-ICSI in previously diagnosed low responder patients.

DETAILED DESCRIPTION:
During controlled ovarian hyperstimulation (COH), most of the early antral follicles are required to grow coordinately. Marked follicular size discrepancies during COH imply that an important number of follicles undergo unsatisfactory maturation. It has been proved that follicular priming with estradiol during the luteal phase of the cycle prior to COH or testosterone treatment during the early follicular phase of the COH cycle may increase the amount of oocytes and embryos retrieved. Nevertheless there are no prospective studies comparing such approaches. The present study consist of two phases:

The present study consists of two different phases:

* Phase I: (Non randomized) Identification of confirmed low responder patients. Potential low responder patients will be subjected to an standardized ovarian hyperstimulation protocol
* Phase II: (Randomized) those patients, once confirmed as low responders, will be offered the opportunity to enter the interventional part of the study, being randomized to three different treatment groups: estradiol, testosterone or combined progestagens and estrogens prior to the IVF-ICSI cycle. The previous cycle (phase I) will be used as a self-control for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1 (Non randomized. The patient must fit the first plus at least other 2 criteria)

   * Infertility requiring an IVF/ICSI treatment
   * Age ≥ 38 years
   * Basal FSH ≥ 10 mUI/ml (day 3 of the cycle)
   * Serum AMH ≤ 5 pmol/l
   * Antral follicular count ≤ 6 (day 3 of the cycle)
2. Phase 2 (Randomized. The patient must fit at least one criterion regarding the day of GNRH analogue administration during the cycle performed in Phase 1)

   * Less than 4 follicles which mean diameter measuring more than 16mm
   * Serum estradiol levels ≤ 500 pg/ml
   * 4 MII or less than 4 MII oocytes retrieved

Exclusion Criteria:

* Patients suffering of endometriosis
* Patients having progesterone levels ≤ 4 ng/ml (day 21 of the cycle)
* Patients having a partner affected by severe oligo/astheno/teratozoospermia

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of MII oocytes retrieved | 36h after GnRH analogue administration

SECONDARY OUTCOMES:
Total number of follicles punctured | 36h after GnRH analogue administration
Total number of oocytes retrieved | 36h after GnRH analogue administration
Total number of viable embryos | 48h after follicular puncture
Serum and Follicular hormonal levels (testosterone, androstenedione, estradiol) | 36h after GnRH analogue administration
Granulosa cells genetic expression profile | 36h after GnRH analogue administration
Implantation rate | 15 days after embryo transfer
Pregnancy rate | 15 days after embryo transfer
Clinical pregnancy rate | 5 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: César Díaz, M.D., Principal Investigator — La Fe University Hospital. Department of Obstetrics and Gynecology; Antonio Pellicer, Professor, Study Director — La Fe University Hospital. Department of Obstetrics and Gynecology; Alicia Marzal, M.D., Study Chair — La Fe University Hospital. Department of Obstetrics and Gynecology
Locations (1):
- La Fe University Hospital. Department of Obstetrics and Gynecology, Valencia, Spain

REFERENCES:
- [Background] Fanchin R, Salomon L, Castelo-Branco A, Olivennes F, Frydman N, Frydman R. Luteal estradiol pre-treatment coordinates follicular growth during controlled ovarian hyperstimulation with GnRH antagonists. Hum Reprod. 2003 Dec;18(12):2698-703. doi: 10.1093/humrep/deg516. PMID 14645194
- [Background] Fabregues F, Penarrubia J, Creus M, Manau D, Casals G, Carmona F, Balasch J. Transdermal testosterone may improve ovarian response to gonadotrophins in low-responder IVF patients: a randomized, clinical trial. Hum Reprod. 2009 Feb;24(2):349-59. doi: 10.1093/humrep/den428. Epub 2008 Dec 3. PMID 19054777
- [Derived] Escriva AM, Diaz-Garcia C, Monterde M, Rubio JM, Pellicer A. Antral Follicle Priming Before Intracytoplasmic Sperm Injection in Previously Diagnosed Low Responders: A Randomized Controlled Trial (FOLLPRIM). J Clin Endocrinol Metab. 2015 Jul;100(7):2597-605. doi: 10.1210/jc.2015-1194. Epub 2015 May 8. PMID 25955224